CLINICAL TRIAL: NCT04635540
Title: A Pilot Study Assessing the Benefits of a Dementia Caregiver Educational Brochure on Decreased Empathy and Emotion Recognition in Patients With Neurodegenerative Disease
Brief Title: Decreased Empathy and Emotion Recognition in Patients With Neurodegenerative Disease
Acronym: Empathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-6350
Record Dates: First submitted 2020-03-30; First posted 2020-11-19 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Neuro-Degenerative Disease; Dementia; Caregiver Burnout; Alzheimer Disease; Frontotemporal Lobar Degeneration; Parkinson Disease; Vascular Dementia
MeSH Terms: conditions — Dementia; Caregiver Burden; Alzheimer Disease; Frontotemporal Lobar Degeneration; Parkinson Disease; Dementia, Vascular

STUDY DESIGN:
Intervention Model Description: Every caregiver and patient dyad will complete the study tasks. The caregiver will receive a 1 month follow up call.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental): The Interventional Arm will receive the educational brochure and complete the study tasks and questionnaires.
  Interventions: Behavioral: Educational Brochure

INTERVENTIONS:
Behavioral: Educational Brochure — Educational brochure on decreased empathy and emotion recognition in patients with neurodegenerative disease

SUMMARY:
This study evaluates an educational brochure tailored to caregivers of people with Alzheimer's disease, Parkinson's disease dementia, Lewy body disease, frontotemporal dementia, and vascular disease dementia. The goal of the brochure is educating caregivers about the decreased ability to detect emotion and decreased empathy that can be seen in dementia, increasing caregiver competence in providing care, and teaching caregivers ways to manage over time that lessens burden and improves quality of life.

DETAILED DESCRIPTION:
The 1.5-hour initial visit will involve the caregiver completing questionnaires, structured interviews, and a computer task, and the person with dementia completing a computer task. A 20-30 minute follow-up phone call with the caregiver one month after the initial visit will involve completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* All caregivers who visit the UHN Memory Clinic with a patient with a neurodegenerative disease will be asked to participate.
* The patient must be aged 50 to 95 (inclusive) and speak English
* The caregiver must be aged 30 to 95 (inclusive) and speak English.
* The patients must have a diagnosis of one of the following conditions: Alzheimer's Disease, Parkinson's Disease/Dementia with Lewy Body, Frontotemporal Lobar Degeneration-syndromes or Vascular Dementia.
* The patient must have a Montreal Cognitive Assessment (MOCA) score of 10-25

Exclusion Criteria:

* Not English speaking.
* Patients who do not have a caregiver that would be able to participate in the study.
* Caregivers who do not have a patient being followed at the UHN Memory Clinic

Ages: 30 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Abbreviated form of the Emotion Evaluation Test (EET) from The Awareness of Social Inference Test (TASIT) | Baseline Visit
  Subjects watch brief (∼ 20s) videos of actors performing semantically neutral scripts portraying one of the seven basic emotions (happy, surprised, neutral, sad, anxious, frightened, revolted), and must choose the correct emotion. The maximum score is 14 and lower scores on this test indicate greater impairment in emotion recognition. Patients and caregivers will be tested separately in a quiet room. No feedback is provided after each clip. Caregivers will be asked to predict the patient's response after each clip. A caregiver accuracy score will be computed by subtracting the patient's actual TASIT-EET score and the caregiver's predicted TASIT-EET score.
Value of educational material | Baseline Visit
  The caregivers will rate the brochure's quality by answering a 7-item questionnaire. The maximum score is 35, with higher scores indicating better quality and helpfulness of the educational brochure.
Change in understanding before and after reading the educational material | Baseline Visit and 1 month after the Baseline visit
  The caregivers will rate their understanding of decreased empathy and emotion recognition changes in people with neurodegenerative disease by answering a 5-item questionnaire. The maximum score is 25 and higher scores will indicate that the caregiver perceives the patient as capable of recognizing the emotions of other people very well.
Caregiver empathy assessment of patient | Baseline Visit
  Empathy will be evaluated using the Interpersonal Reactivity Index (IRI), which measures both the cognitive and emotional aspects of empathy. Informants fill out a 28-item self report questionnaire describing the subject's current characteristics. Scores range from 28-140. Higher scores indicate better performance.
Caregiver functional assessment of patient | Baseline Visit
  Functional capacity will be evaluated with the Functional Activities Questionnaire (FAQ). Informants fill out a 10-item questionnaire describing the patient's current functional capacity. Scores range from 0-30 with a cut-off score of 9 indicating impaired function and possible cognitive impairment.
Caregiver neuropsychiatric assessment of patient | Baseline Visit
  The neuropsychiatric inventory (NPI) will be administered to caregivers to assess neuropsychiatric symptoms (NPS) in individuals with dementia. The NPI assesses the presence of the following NPS over the period of four weeks: delusions, hallucinations, agitation, depression/dysphoria, anxiety, euphoria/elation, apathy indifference, disinhibition, irritability/lability, aberrant motor behaviour, sleep, and appetite and eating disorder. Caregivers are asked about the frequency (4-point scale) and severity (3-point scale) of these symptoms and on caregiver distress. A total score for each symptom is obtained by multiplying the frequency and severity score, giving a maximum score of 144 with higher scores reflecting increased frequency and severity of NPS. Lastly, caregiver distress is rated on a 6-point scale.
Caregiver staging of dementia severity assessment of patient | Baseline Visit
  The Clinical Dementia Rating Scale (CDR) modified version assesses 8 domains of global dementia using a five-point scale, including: memory, orientation, judgment/problem solving, community affairs, home and hobbies, personal care, behavioural comportment and personality, and language. It is used as a staging scale to assess the severity of dementia. It is performed through a semi-structured analysis with a caregiver. The CDR sum of boxes will be used in the analysis. The maximum sum of boxes is 24 with higher scores showing increased impairment.
Change in caregiver burden at 1 month | Baseline Visit and 1 month after the Baseline Visit
  The Zarit Burden Inventory (ZBI) assesses caregiver burden in individuals caring for patients with dementia. The caregivers filled out a 22-item ZBI questionnaire to evaluate the amount of stress experienced by them due to the person's dementia. Each item is rated on a 5-point scale, and a total score is calculated by taking the sum of individual statements. The score ranges from 0-88 and higher scores on the ZBI indicates increased burden. The change in score from the initial appointment and 1 month follow up will be used in analysis.
Change in caregiver mood symptoms at 1 month | Baseline Visit and 1 month after the Baseline Visit
  The Geriatric Depression Scale (GDS) assesses mood and depression in geriatric patients and will be used for caregivers 50 years old and above. Scores range from 0-15 with higher scores indicating greater symptoms of depression. The Depression Anxiety Stress Scale (DASS) assesses depression, anxiety, and stress and can be used in adults and geriatric patients. The DASS will be used for all caregivers aged 30 years and above. Scores range from 0-63 with higher scores indicating increased symptoms of depression. The change in score from the initial appointment and 1 month follow up will be used in analysis.
Change in caregiver quality of life at 1 month | Baseline Visit and 1 month after the Baseline Visit
  The World Health Organization Quality of Life (WHOQOL-BREF) is a 26-item, self-reported quality of life measure, which measures quality of life in four domains: physical health, psychological health, social relationships, and environment. Answers are rated on a scale of 1-5, where numbers can be in order of increasing satisfaction or decreasing satisfaction depending on the domain and questionnaire item. The score range is from 26-130 with higher scores indicating increased quality of life satisfaction. The change in score from the initial appointment and 1 month follow up will be used in analysis.

SECONDARY OUTCOMES:
Recruitment Rate | through study completion, an average of 1 year
  Number of individuals signing consent/number of individuals approached
Retention Rate | through study completion, an average of 1 year
  Number of those who remain in study/number of participants who have signed consent at the beginning of the study
Completion Rate | through study completion, an average of 1 year
  Number of dyads with completed questionnaire/total subject population (For a questionnaire to be complete, every question must be answered).

CONTACTS AND LOCATIONS:
Overall Officials: Carmela Tartaglia, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form: Patient Consent Form (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT04635540/ICF_000.pdf
  • Informed Consent Form: Caregiver Consent Form (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT04635540/ICF_001.pdf